CLINICAL TRIAL: NCT03651817
Title: Lung Protection Strategy in Open Heart Surgery: Which Tidal Volume is Better 8ml/kg or 6ml/kg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tülay Çardaközü, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KÜ GOKAEK 2018/68
Record Dates: First submitted 2018-07-27; First posted 2018-08-29 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Lung Injury, Acute; Ventilator-Induced Lung Injury; Ventilator Adverse Event
MeSH Terms: conditions — Acute Lung Injury; Ventilator-Induced Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6ml/kg volume (Active Comparator): Patients ventilation will provided with a tidal volume of 6ml/kg
  Interventions: Device: Mechanical ventilation
- 8ml/kg volume (Active Comparator): Patients ventilation will provided with a tidal volume of 8ml/kg
  Interventions: Device: Mechanical ventilation

INTERVENTIONS:
Device: Mechanical ventilation — Patients will be ventilated with anesthesia machine according to the group they belong to

SUMMARY:
Respiratory complications range from 8% to 79% of the frequency after open heart surgery where the patient is on-pump operated by cardiopulmonary machine. There were many changes in physiology due to anesthesia and cardiac surgery which cause volume and barotrauma complications with mechanical ventilation. These complications increase cost by prolonging morbidity and morbidity as well as hospital stay. Intraoperative and postoperative mechanical ventilation strategies can prevent these complications. CPB stimulates the systemic inflammatory response to the secretion of neutrophil, endotoxin and proinflammatory cytokines in the complex, increasing the permeability of the capillaries. Although coronary artery bypass graft surgery (CABG) is associated with a 0.4% to 2.0% acute respiratory distress syndrome (ARDS), mortality is quite high. Lung-protective ventilation strategies commonly used for prevention of ARDS. Ferrando et al. have proposed pulmonary ventilation with a tidal volume (TV) of less than 10 mL / kg as a pulmonary intraoperative protective ventilation strategy. Investigators aimed to compare oxygenation and ventilation parameters with respiratory mechanics in patients who underwent open heart surgery and were ventilated with 6 ml / kg tidal volume and 8 ml / kg TV, which were recommended as lung protective ventilation strategies during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Cardiopulmonary bypass

Exclusion Criteria:

* Severe COPD
* Chronic Anemia
* Active Smoker
* Chronic kidney Disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Change of arterial carbondiokside pressure levels | from the beginning of operation to 6th hour of post-extubation
  Investigators will compare the changes in arterial carbondiokside levels in arterial blood gas samples

SECONDARY OUTCOMES:
Changes in respiratory parameters | from the beginning of the operation to the end of the surgery
  airway pressures will be continuously assessed
Changes in Invasive blood pressures | from the beginning of the operation to the end of the surgery
  Blood pressure will be continuously recorded and assessed due to time intervals
Changes in heart rate | from the beginning of the operation to the end of the surgery
  Heart rate will be continuously recorded and assessed due to time intervals
Changes in central venous pressure | from the beginning of the operation to the end of the surgery
  Continous central venous pressure will ve recorded and assessed due to time intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)